CLINICAL TRIAL: NCT03126279
Title: Predicting Chronic Post TKR Pain by Assessing Central Sensitisation Using Functional Brain MRI
Brief Title: fMRI and Central Sensitization in Chronic Knee Osteoarthritis. A Pre and Post TKR Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Nottingham (Other)
Collaborators: Aalborg University (Other); Medical Research Council (Other Government); Arthritis Research UK (Other); Royal College of Surgeons of Edinburgh (Other)
Responsible Party: Sponsor
Other Study IDs: 10093
Record Dates: First submitted 2017-04-11; First posted 2017-04-24 (Actual); Last update posted 2017-04-24 (Actual); Status verified 2017-04

CONDITIONS: Osteoarthritis; Pain; Postoperative Pain; Surgery
Keywords: Osteoarthritis; Pain; Postoperative Pain
MeSH Terms: conditions — Osteoarthritis; Pain; Pain, Postoperative

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Preoperative Chronic Knee OA Patients: Patients will be recruited from orthopaedic preoperative clinics from those awaiting total knee replacement surgery.
  Interventions: Procedure: Total Knee Replacement Surgery
- Healthy Volunteers: Healthy volunteers will be recruited that are aged match to our OA patient cohort so meaningful comparisons regarding brain activity and pain sensitisation characteristics can be assessed.

INTERVENTIONS:
Procedure: Total Knee Replacement Surgery — All chronic knee osteoarthritis patients will be recruited as they are on the NHS waiting list for a total knee replacement. Only this group will undergo the procedure
  Other Names: Total
  Groups: Preoperative Chronic Knee OA Patients

SUMMARY:
Painful osteoarthritis (OA) is the 4th largest cause of disability in the UK. Preoperative temporal summation, a measure of central pain facilitation, has been shown to predict postoperative pain after total knee replacement surgery (TKR). The assessment of the brain's response to noxious stimuli using non-invasive functional MRI (fMRI) may be key in identifying imaging biomarkers within the brain that map central sensitization changes seen in OA. fMRI may help explain why up to 20% of patients undergoing TKR surgery develop persistent post-operative pain. To test these concepts the study aims to functionally characterise the brain activity related to temporal summation of pain in healthy individuals and OA patients using a novel fMRI cuff algometer. Assessment of outcomes in terms of pain and function will be performed 6 months post TKR surgery

ELIGIBILITY:
Inclusion Criteria:

* OA Group

Unilateral Knee OA No previous knee surgery Able to give informed consent Age > 40 years

- Healthy Volunteers Group

No OA or knee pain Able to give informed consent Age > 40 years

Exclusion Criteria:

-OA Group

Major medical, psychiatric, neurological Cx Other chronic pain condition (fibromyalgia) Contraindications to MRI Active Cancer Neuropathic drug treatment

-Healthy Volunteers Group

Pregnancy Lower limb pain or previous knee surgery Contraindications to MRI Active Cancer Major medical, psychiatric, neurological condition

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with predominelaty unilateral knee osteoarthritis awaiting for total knee replacement surgery for pain will be included. Patients will recruited from Nottingham University Hospitals NHS Trust. Healthy volunteers will also be recruited as part of this study and they will be recruited from posters and advertisement within the university.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2015-08; Primary Completion 2017-06 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Brain activity related to temporal summation of pain in healthy individuals and OA patients using a novel fMRI cuff algometer. | 6 months post total knee replacement surgery
  Using BOLD fMRI we aim to assess the difference in neural brain activity between patients with chronic knee OA pain and a group of healthy volunteers and to assess the reversal of this activity pattern 6 months post TKR surgery

SECONDARY OUTCOMES:
Assessment of knee pain using the Visual Analogue Scale for Pain (0-10) | 6 months post total knee replacement surgery
  Pain using visual analogue scale
Assessment of improvement in the Oxford Knee Score | 6 months post total knee replacement surgery
  pain and function outcome measure
Assessment of change in healthy related quality of life measure using the EQ5D-5L questionnaire | 6 months post total knee replacement
  quality of life index measure

CONTACTS AND LOCATIONS:
Overall Officials: Dorothee P Auer, PhD, Principal Investigator — The University of Nottingham
Locations (1):
- Academic Division of Trauma, Orthopaedics and Sports Medicine, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No